CLINICAL TRIAL: NCT01304277
Title: A Phase II Comparability Study Between Replagal® Produced From Agalsidase Alfa Manufactured by 2 Different Processes in Adult Male Patients With Fabry Disease
Brief Title: This Study is Designed to Evaluate PD/PK and Safety of Replagal Manufactured by Two Different Processes.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HGT-REP-082
Record Dates: First submitted 2011-02-15; First posted 2011-02-25 (Estimated); Results first posted 2014-04-25 (Estimated); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Fabry Disease
Keywords: Replagal
MeSH Terms: conditions — Fabry Disease | interventions — agalsidase alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Replagal® (0.2 mg/kg, IV, EOW) (Experimental): Screening period of approximately 14 days during which all patients received 1 infusion of 0.2 mg/kg Replagal RB (Week 0)
  Treatment period of 14 weeks during which all patients received 7 infusions of 0.2 mg/kg Replagal AF
  Interventions: Biological: agalsidase alfa

INTERVENTIONS:
Biological: agalsidase alfa
  Other Names: Replagal

SUMMARY:
This study is designed to evaluate safety and PK/PD in Canadian Fabry patients.

DETAILED DESCRIPTION:
In 2008, a change in the agalsidase alfa drug substance manufacturing process was made. There are no changes to the drug product formulation, manufacturing site, manufacturing process, or container closure.

An agalsidase alfa bioreactor manufacturing process (agalAF1) utilizing animal component-free media replaced the previous roller bottle (RB) process.

This study is designed to provide PD/PK and safety data. The assessment schedule is designed to capture the PK profile of drug uptake in the blood as well the pharmacologic effect which manifests over the course of weeks. Each patient will serve as his own control.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must be diagnosed with Fabry disease using the following criteria: The patient is a hemizygous male with Fabry disease as confirmed by a deficiency of α-galactosidase A activity measured in serum, leukocytes, or fibroblasts or has a confirmed mutation of the α-galactosidase A gene.
2. Patient is male and between 18 and 65 years of age, inclusive.
3. Patient must be willing to remain in the clinic as required by the study and comply with the procedures and evaluations of the study.
4. At the time of confirmation of study eligibility visit, patients must have received at least 26 weeks of treatment with RB Replagal at a dose of 0.2 mg/kg administered IV EOW.
5. Patient provides informed consent.

Patients who are naive to ERT:

1. Treatment naive patients must have a pretreatment plasma Gb3 level above the normal range (if value is available).

Exclusion Criteria:

1. Patient is unable to be venipunctured and/or tolerate venous access.
2. Patient has tested positive for anti-agalsidase alfa antibodies either at screening or confirmation of eligibility visit.
3. Patient had pre-ERT plasma Gb3 levels within the normal range (if value is available).
4. Patient is participating in any other Shire HGT investigational study.
5. Patient is currently on dialysis, is expected to begin dialysis during the study, has received a kidney transplant, or is on the renal transplant waiting list.
6. Patient is unable to comply with the protocol (eg, clinical relevant medical condition making implementation of the protocol difficult, unstable social situation, or otherwise unlikely to complete the study) or is, in the opinion of the Investigator, otherwise unsuited for the study.
7. The patient is enrolled in another clinical study that involves clinical investigations or use of any investigational product (drug or device), except for the Canadian Fabry Disease Initiative, within 6 months prior to receiving the first dose of AF Replagal in this study or at any time during the study.
8. The patient has previously received AF Replagal prior to study entry.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2011-11-17 (Actual); Primary Completion 2012-12-28 (Actual); Study Completion 2012-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (5):
- Canada (5):
  - University of Alberta Hospital, Edmonton, Alberta
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - The Hospital for Sick Children, Toronto, Ontario
  - INC Research, Toronto, Ontario
  - Hopital du Sacre-Coeur de Montreal, Montreal, Quebec

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient participated in the study on 06 December 2011 and the last patient completed the study procedures on 28 December 2012.
Groups:
- Replagal® (0.2 mg/kg, EOW): Patients who had received Replagal RB for at least 26 weeks prior to entering the study REP-082, received 1 dose of Replagal RB at baseline before switching to Replagal AF. They then received 14 weeks of treatment with Replagal AF.
Period: Screening (Replagal RB, Week 0- Week 2)
Arm/Group | Replagal® (0.2 mg/kg, EOW)
Started | 17
Completed | 17
Not Completed | 0
Period: Treatment (Replagal AF, Week 2- EOS)
Arm/Group | Replagal® (0.2 mg/kg, EOW)
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Replagal® (0.2 mg/kg, EOW)
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.8 (13.589)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 17
Region of Enrollment [Count of Participants; unit: Participants]
  CANADA | 17
Study Specific Characteristic [Urine Gb3] [Mean (Standard Deviation); unit: nmol/g creatinine] — Baseline is the average of Gb3 (globotriaosylceramide) levels on RB Replagal at screening, Week 0, and Week 2 prior to AF Replagal dosing.
  nmol/g creatinine | 919.27 (990.144)
Study Specific Characteristic [Plasma Gb3] [Mean (Standard Deviation); unit: nmol/mL] — Baseline is the average of Gb3 (globotriaosylceramide) levels on RB Replagal at screening, Week 0, and Week 2 prior to AF Replagal dosing.
  nmol/mL | 5.276 (1.562)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 16 (EOS) in Urine Gb3 Levels
Time Frame: Baseline to EOS
Measure: Mean (Standard Deviation); unit: (nmol/g creatinine)
Arm/Group | Replagal® (0.2 mg/kg, EOW)
Number analyzed (Participants) | 17
(nmol/g creatinine) | -28.68 (192.659)

2. Secondary Outcome: Change From Baseline to Week 16 (EOS) in Plasma Gb3 Levels
Time Frame: Baseline to EOS
Measure: Mean (Standard Deviation); unit: (nmol/mL)
Arm/Group | Replagal® (0.2 mg/kg, EOW)
Number analyzed (Participants) | 17
(nmol/mL) | 0.170 (0.503)

3. Secondary Outcome: Dose-normalized Area Under the Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Sample (AUClast/Dose)
Description: The dose-normalized calculation was performed by dividing the pharmacokinetic parameter by the administered dose.
Time Frame: Week 0 to Week 14
Measure: Geometric Mean (90% Confidence Interval); unit: Ratio
Arm/Group | Replagal® (0.2 mg/kg, EOW)
Number analyzed (Participants) | 17
Ratio
  Week 14 versus 0 | 0.65 [0.61 to 0.72]
  Week 14 versus 2 | 1.05 [0.94 to 1.23]

4. Secondary Outcome: Dose-normalized AUC Extrapolated to Infinity (AUC∞/Dose)
Description: The dose-normalized calculation was performed by dividing the pharmacokinetic parameter by the administered dose.
Time Frame: Week 0 to Week 14
Measure: Geometric Mean (90% Confidence Interval); unit: Ratio
Arm/Group | Replagal® (0.2 mg/kg, EOW)
Number analyzed (Participants) | 17
Ratio
  Week 14 versus 0 | 0.67 [0.62 to 0.75]
  Week 14 versus 2 | 1.07 [0.97 to 1.26]

5. Secondary Outcome: Dose-normalized Maximum Serum Concentration (Cmax/Dose)
Description: The dose-normalized calculation was performed by dividing the pharmacokinetic parameter by the administered dose.
Time Frame: Week 0 to Week 14
Measure: Geometric Mean (90% Confidence Interval); unit: Ratio
Arm/Group | Replagal® (0.2 mg/kg, EOW)
Number analyzed (Participants) | 17
Ratio
  Week 14 versus 0 | 0.81 [0.76 to 0.91]
  Week 14 versus 2 | 1.05 [0.96 to 1.21]

6. Secondary Outcome: To Assess Safety and Tolerability by Anti-agalsidase Alfa Antibody Status (in Serum) at End of Study
Time Frame: EOS
Measure: Number; unit: participants
Arm/Group | Replagal® (0.2 mg/kg, EOW)
Number analyzed (Participants) | 17
participants
  Anti-Agalsidase alfa Antibody Negative | 13
  Anti-Agalsidase alfa Antibody Positive (IgG) | 2
  Anti-Agalsidase alfa Antibody Positive (IgM) | 2

7. Secondary Outcome: Overall Summary of TEAEs by Treatment (Replagal RB and Replagal AF)
Description: To Assess Safety and Tolerability by Anti-agalsidase Alfa Antibody Status, concomitant medication, vital signs and ECG.
Time Frame: Week 2 to EOS
Measure: Number; unit: participants
Groups:
- Replagal RB: Patients who had received Replagal RB for at least 26 weeks prior to entering the study REP-082.
- Replagal AF: Patients received 7 EOW infusions of treatment with Replagal AF from week 2 to week 14 in REP-082.
- Overall: Overall number of patients who experienced adverse events during the course of REP-082 study.
Arm/Group | Replagal RB | Replagal AF | Overall
Number analyzed (Participants) | 17 | 17 | 17
participants
  No TEAE | 9 | 5 | 5
  Experienced at least one TEAE | 8 | 12 | 12
  Deaths | 0 | 0 | 0
  Discontinued due to a TEAE | 0 | 0 | 0
  Experienced at least one drug-related TEAE | 3 | 3 | 3
  Experienced at least one SAE | 0 | 2 | 2
  At least one severe or life- threatening TEAE | 1 | 1 | 1
  At least one IRR (infusion related reaction) | 1 | 1 | 1

ADVERSE EVENTS:
Time Frame: Baseline to EOS
Groups:
- Replagal® (0.2 mg/kg, IV, EOW): Overall patients that participated in REP-082
Arm/Group | Replagal® (0.2 mg/kg, IV, EOW)
Serious Adverse Events (participants affected / at risk) | 2/17
Other Adverse Events (participants affected / at risk) | 12/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Replagal® (0.2 mg/kg, IV, EOW) (N=17)
Cardiac arrest (Cardiac disorders) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Replagal® (0.2 mg/kg, IV, EOW) (N=17)
Bradycardia (Cardiac disorders) | 1 (1)
Visual impairment (Eye disorders) | 1 (2)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (4)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (5)
Nausea (Gastrointestinal disorders) | 2 (5)
Vomiting (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 3 (3)
Oedema peripheral (General disorders) | 2 (3)
Pyrexia (General disorders) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (3)
Upper respiratory tract infection (Infections and infestations) | 2 (3)
Excoriation (Injury, poisoning and procedural complications) | 1 (1)
Joint sprain (Injury, poisoning and procedural complications) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1)
Blood potassium decreased (Investigations) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (5)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (5)
Headache (Nervous system disorders) | 2 (4)
Migraine (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 2 (7)
Depression (Psychiatric disorders) | 1 (1)
Stress (Psychiatric disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Gynaecomastia (Reproductive system and breast disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Shire's agreements with investigators vary. All agreements provide Shire the right to embargo communications regarding trial results prior to public release for a period ≤180 days from the time submitted to Shire for review. Shire does not prohibit publication, but can require the removal of confidential information (excluding trial results) and can request postponement of a single-center publication until after disclosure of the trial's multi-center publication.